CLINICAL TRIAL: NCT03034655
Title: Reducing Rate of Falls in Older People With the Improvement of Balance by Means of Vestibular Rehabilitation (ReFOVeRe Study): Optimizing Costs
Brief Title: Reducing Rate of Falls in Older People by Means of Vestibular Rehabilitation (ReFOVeRe Study)
Acronym: ReFOVeRe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Andrés Soto-Varela, Professor and Attending Physician, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI1500329
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Dizziness Chronic; Fall
Keywords: Vestibular rehabilitation; Falls in elderly; Computerized dynamic posturography; Mobile posturography

STUDY DESIGN:
Intervention Model Description: Experimental study, single-center, open, randomized (balanced blocks of patients) in four branches in parallel, in 220 elderly patients (over 65 years) with high risk of falls; follow-up period: twelve months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: After the first screening visit, the patients who grant their consent will be included in the study and randomised to one of the following study arms. Randomisation will be performed by C.H.U de Santiago Clinical Epidemiology and Biostatistics Unit. Once the informed consent form is signed, the care provider will contact the unit, which will give him the code of the arm to which the patient is assigned. A n= 20 block balanced randomisation sequence will be used. The investigator will analyse results and evolution, being blind type and duration of vestibular rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CDP exercises (10 sessions) (Experimental): Group A. The Smart Equitest program was used with a protocol of 10 exercises per session, which were customized depending on each patient´s deficit. The exercises involve visual biofeedback together with sensitive, real-time monitoring of movement. In some exercises, patients must maintain their center of gravity (COG) over the base of support, while in others the COG must be moved to a series of targets. In addition, the support surface and/or visual surround may also move in response to the patient´s own movement. The exercise difficulty was progressively increased throughout the rehabilitation sessions. The duration of each session was approximately 15 minutes. The distribution of sessions was one per day and five per week (2 weeks).
  Interventions: Device: CDP; Other: 10 sessions
- CDP exercises (5 sessions) (Experimental): Group B. Same as group A, except for the number of sessions (5) and the distribution of sessions (one daily, every other day, two weeks).
  Interventions: Device: CDP; Other: 5 sessions
- Mobile posturography exercises (10 sess) (Experimental): Group C. Up to six tasks with the most prominent deviations from normative control values were included in the training program. Training was performed by using the training function of Vertiguard1-RT device. This neurofeedback system contains one vibration stimulator on the front, back, left and right side, respectively. Training was performed daily under supervision of a physician over 2 weeks (10 sessions, weekend was excluded). A training session consisted of 5 repetitions of six selected training tasks. The patient received a vibrotactile feedback signal during training in those directions which showed a higher body sway than preset thresholds. Vibration was reinforced with increasing sway No vibrotactile feedback was applied if the patient's sway was below preset thresholds. The exercise difficulty was progressively increase throughout the rehabilitation sessions.
  Interventions: Device: Mobile posturography; Other: 10 sessions
- Mobile posturography exercises (5 sess) (Experimental): Group D. Same as group A, except for the number of sessions (5) and the distribution of sessions (one daily, every other day, two weeks).
  Interventions: Device: Mobile posturography; Other: 5 sessions

INTERVENTIONS:
Device: CDP — Vestibular rehabilitation using CDP
  Other Names: Computerized Dynamic Posturography
  Arms: CDP exercises (10 sessions); CDP exercises (5 sessions)
Device: Mobile posturography — Vestibular rehabilitation using mobile posturography
  Other Names: Vertiguard's Mobile Posturography
  Arms: Mobile posturography exercises (10 sess); Mobile posturography exercises (5 sess)
Other: 10 sessions — Vestibular rehabilitation, ten sessions
  Arms: CDP exercises (10 sessions); Mobile posturography exercises (10 sess)
Other: 5 sessions — Vestibular rehabilitation, five sessions
  Arms: CDP exercises (5 sessions); Mobile posturography exercises (5 sess)

SUMMARY:
The aim of this study is to evaluate and compare the effectiveness of vestibular rehabilitation developed using computerized dynamic posturography or a mobile posturographic system with vibrotactile stimulation, to improve the balance in older people and reduce the number of falls.

DETAILED DESCRIPTION:
Accidental falls, particularly in the elderly, are one of the most important socio-healthcare problems of ageing western societies. Many factors condition and favour falls; one of them is old age, usually related to a decline in sensorial functions and worsening of balance Vestibular rehabilitation has been shown to be effective to improve balance and reduce the number of falls in older people. Previous studies have demonstrated that exercises in computerized dynamic posturography (CDP) are more effective than other vestibular rehabilitation strategies in this group of age. But CDP is very expensive and not widespread. It would be important to minimize cost of posturographic vestibular rehabilitation.

This study compare vestibular rehabilitation with two different posturographic devices (CDP and mobile posturographic system with vibrotactile stimulation), in people over 65 years. Additionally, we try to assess whether the reduction in the number of vestibular rehabilitation sessions (five) leads to an improvement in balance and in reducing the number of falls similar to those obtained with ten sessions.

ELIGIBILITY:
Inclusion Criteria:

Persons with a high risk of falling shall meet at least two of the following requirements:

* Having fallen at least once in the last 12 months.
* Using more than 15 seconds or needing support in the TUG test.
* Obtaining a mean CDP SOT balance score of < 68%.
* Having fallen at least once in the CDP SOT.
* A score in Mobile posturography gSBDT > 60 %.

Exclusion Criteria:

* Cognitive decline or reduce cultural level that prevents the patient from understanding the assessment, vestibular rehabilitation exercises and granting informed consent.
* Organic conditions that prevent standing on two feet, necessary for assessment of balance and performance of VR exercises.
* Balance disorders caused by conditions other than age (neurologic, vestibular,....).
* Current treatment with drugs that potentially disturb balance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
CDP Average | 12 months
  Average score in the Sensory Organization Test of the Computerized Dynamic Posturography

SECONDARY OUTCOMES:
Mobile posturografphy gSBDT | 12 months
  Geriatric Standard Balance Deficit Test (gSBDT) score in mobile posturography
Falls | 12 months
  Number of falls after vestibular rehabilitation
DHI | 12 months
  Dizziness Handicap Inventory score; it assesses disability perceived by the patient in relation to instability
Short FES-I | 12 months
  Score of a shortened version of the falls efficacy scale-international to assess fear of falling
TUG | 12 months
  Timed up and go test: time (in seconds), number of steps and need for support

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Soto-Varela, PhD, Principal Investigator — Hospital Clinico Universitario de Santiago
Locations (1):
- Complexo Hospitalario Universitario, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soto-Varela A, Rossi-Izquierdo M, Del-Rio-Valeiras M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Santos-Perez S. Vestibular rehabilitation with mobile posturography as a "low-cost" alternative to vestibular rehabilitation with computerized dynamic posturography, in old people with imbalance: a randomized clinical trial. Aging Clin Exp Res. 2021 Oct;33(10):2807-2819. doi: 10.1007/s40520-021-01813-2. Epub 2021 Mar 7. PMID 33677737
- [Derived] Soto-Varela A, Rossi-Izquierdo M, Del-Rio-Valeiras M, Vaamonde-Sanchez-Andrade I, Faraldo-Garcia A, Lirola-Delgado A, Santos-Perez S. Presbyvestibulopathy, Comorbidities, and Perception of Disability: A Cross-Sectional Study. Front Neurol. 2020 Oct 30;11:582038. doi: 10.3389/fneur.2020.582038. eCollection 2020. PMID 33250848
- [Derived] Soto-Varela A, Rossi-Izquierdo M, Del-Rio-Valeiras M, Vaamonde-Sanchez-Andrade I, Faraldo-Garcia A, Lirola-Delgado A, Santos-Perez S. Vestibular Rehabilitation Using Posturographic System in Elderly Patients with Postural Instability: Can the Number of Sessions Be Reduced? Clin Interv Aging. 2020 Jun 26;15:991-1001. doi: 10.2147/CIA.S263302. eCollection 2020. PMID 32617000
- [Derived] Soto-Varela A, Rossi-Izquierdo M, Del-Rio-Valeiras M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Santos-Perez S. Modified Timed Up and Go Test for Tendency to Fall and Balance Assessment in Elderly Patients With Gait Instability. Front Neurol. 2020 Jun 12;11:543. doi: 10.3389/fneur.2020.00543. eCollection 2020. PMID 32595593
- [Derived] Soto-Varela A, Gayoso-Diz P, Faraldo-Garcia A, Rossi-Izquierdo M, Vaamonde-Sanchez-Andrade I, Del-Rio-Valeiras M, Lirola-Delgado A, Santos-Perez S. Optimising costs in reducing rate of falls in older people with the improvement of balance by means of vestibular rehabilitation (ReFOVeRe study): a randomized controlled trial comparing computerised dynamic posturography vs mobile vibrotactile posturography system. BMC Geriatr. 2019 Jan 3;19(1):1. doi: 10.1186/s12877-018-1019-5. PMID 30606112